CLINICAL TRIAL: NCT02658981
Title: A Phase I Trial of Anti-LAG-3 or Anti-CD137 Alone and in Combination With Anti-PD-1 in Patients With Recurrent GBM
Brief Title: Anti-LAG-3 Alone & in Combination w/ Nivolumab Treating Patients w/ Recurrent GBM (Anti-CD137 Arm Closed 10/16/18)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABTC 1501; IRB00095527 (Other: JHM IRB); UM1CA137443 (NIH)
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Glioblastoma; Gliosarcoma; Recurrent Brain Neoplasm
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — spartalizumab; Nivolumab; urelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- A1 Anti-LAG-3 (Experimental): Patients receive Anti-LAG-3 monoclonal antibody BMS-986016 IV over 60 minutes and on days 1 and 15. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Pharmacological Study
  Laboratory Biomarker Analysis
  Interventions: Biological: Anti-LAG-3 Monoclonal Antibody BMS 986016; Other: Pharmacological Study; Other: Laboratory Biomarker Analysis
- A2 Anti-CD137 (Urelumab) (Experimental): Patients receive Anti-CD137 (Urelumab) IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 15 courses in the absence of disease progression or unacceptable toxicity
  Pharmacological Study
  Laboratory Biomarker Analysis
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Anti-CD137
- B1 Anti-LAG3 + Anti-PD-1 (nivolumab) (Experimental): Patients receive Anti-PD-1 (nivolumab) IV over 60 minutes and anti-LAG-3 monoclonal antibody BMS-986016 IV on days 1 and 15. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Pharmacological Study
  Laboratory Biomarker Analysis
  Interventions: Biological: Anti-LAG-3 Monoclonal Antibody BMS 986016; Biological: Anti-PD-1; Other: Laboratory Biomarker Analysis
- B2 Anti-CD137 + Anti-PD-1 (Experimental): Patients receive Anti-PD-1 (nivolumab) IV over 60 minutes on days 1 and 15 and Anti-CD137 (urelumab) IV on day 1. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  (2pts enrolled before the Anti-CD137 antibody (BMS-663513 - urelumab) treatment arm closed by BMS on 10/16/18 due to closure of BMS Urelumab development program. Subjects currently on treatment may continue.)
  Pharmacological Study
  Laboratory Biomarker Analysis
  Interventions: Biological: Anti-PD-1; Other: Pharmacological Study; Other: Laboratory Biomarker Analysis; Biological: Anti-CD137
- Intratumoral Studies (Experimental): Patients pre-operatively receive either anti-LAG-3 monoclonal antibody BMS-986016 (Arm A1), or urelumab (Arm A2), or nivolumab and anti-LAG-3 monoclonal antibody BMS-986016 as in Part B (B1)), or nivolumab and urelumab as in Part B (B2). Within 45 days of surgical resection, patients post-operatively receive drug from one of the four arms.
  (3pts enrolled before the Anti-CD137 antibody (BMS-663513 - urelumab) treatment arm closed by BMS on 10/16/18 due to closure of BMS Urelumab development program. Subjects currently on treatment may continue.)
  Interventions: Biological: Anti-LAG-3 Monoclonal Antibody BMS 986016; Biological: Anti-PD-1; Other: Pharmacological Study; Other: Laboratory Biomarker Analysis; Biological: Anti-CD137

INTERVENTIONS:
Biological: Anti-LAG-3 Monoclonal Antibody BMS 986016 — Given IV
  Arms: A1 Anti-LAG-3; B1 Anti-LAG3 + Anti-PD-1 (nivolumab); Intratumoral Studies
Biological: Anti-PD-1 — Given IV
  Other Names: BMS-936558; Nivolumab
  Arms: B1 Anti-LAG3 + Anti-PD-1 (nivolumab); B2 Anti-CD137 + Anti-PD-1; Intratumoral Studies
Other: Pharmacological Study — Correlative Studies
  Arms: A1 Anti-LAG-3; B2 Anti-CD137 + Anti-PD-1; Intratumoral Studies
Other: Laboratory Biomarker Analysis — Correlative Studies
Biological: Anti-CD137 — Given IV
  Other Names: urelumab
  Arms: A2 Anti-CD137 (Urelumab); B2 Anti-CD137 + Anti-PD-1; Intratumoral Studies

SUMMARY:
This phase I trial studies the safety and best dose of anti-LAG-3 (anti-LAG-3 monoclonal antibody BMS-986016) or urelumab alone and in combination with nivolumab in treating patients with glioblastoma that has returned (recurrent). Anti-LAG-3 monoclonal antibody BMS-986016, urelumab, and nivolumab are antibodies (a type of protein) that may stimulate the cells in the immune system to attack tumor cells. It is not yet known whether anti-LAG-3 monoclonal antibody BMS-986016 or urelumab alone or in combination with nivolumab may kill more tumor cells. (The Anti-CD137 antibody (BMS-663513 - urelumab) treatment arm closed by BMS on 10/16/18 due to closure of BMS Urelumab development program. Subjects currently on treatment may continue.)

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine a maximum tolerated dose or maximum administrated dose of anti-lymphocyte activation gene-3 (LAG-3) antibody (BMS-986016) (anti-LAG-3 monoclonal antibody BMS-986016) and anti-cluster of differentiation 137 (CD137) antibody (BMS- 663513) (urelumab) given independently and in combination with anti-programmed death-1 (PD-1) antibody (nivolumab, BMS-936558) safely in patients with recurrent glioblastoma multiforme (GBM).

SECONDARY OBJECTIVES:

I. To estimate overall survival. II. To estimate 1 year progression-free survival (PFS) rate. III. To estimate radiographic response (radiographic assessment in neuro-oncology [RANO] and immunotherapy response assessment for neuro-oncology [iRANO]).

TERTIARY OBJECTIVES:

I. To assess the pharmacodynamic effects of anti-LAG-3 antibody (BMS-986016), anti-CD137 antibody (BMS- 663513), and/or anti-PD-1 antibody (BMS-936558) on biomarkers in peripheral blood, including the T cell compartments, and serum proteins (cytokines and other immune modulators).

II. To assess the pharmacodynamic activity in tumor tissue and peripheral blood in treated subjects who undergo optional tumor biopsies.

III. To explore potential associations between biomarker measures and anti-tumor activity by analyzing markers of inflammation, immune activation, host tumor growth factors, and tumor-derived proteins in the pre-treatment and on-treatment setting.

IV. To further characterize the occupancy and immune cell function at multiple dose levels of anti-LAG-3 antibody (BMS-986016), anti-CD137 antibody (BMS-663513), and/or anti-PD-1 antibody (BMS-936558).

V. To explore characteristics of tumor immune microenvironment changes after the treatment of anti-LAG-3, anti-CD137, and its combination treatment with anti- PD-1 in surgically indicated patients undergoing tumor resection

OUTLINE:

PART A: This is a dose-escalation study of the monotherapy of Anti-LAG-3 monoclonal antibody BMS-986016 and Anti-CD137 (urelumab). Patients are assigned to 1 of 2 arms.

ARM I: Patients receive anti-LAG-3 monoclonal antibody BMS-986016 intravenously (IV) on days 1 and 15. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive anti-CD137 (urelumab) IV on day 1. Treatment repeats every 21 days for up to 15 courses in the absence of disease progression or unacceptable toxicity.

PART B: This is the dose-escalation combination therapy portion study of Anti-LAG-3 monoclonal antibody BMS-986016 plus Anti-PD-1(nivolumab) and Anti-CD137 (urelumab) plus Anti-PD-1 (nivolumab). Patients are assigned to 1 of 2 arms.

ARM I: Patients receive Anti-PD-1 (nivolumab) IV over 60 minutes and anti-LAG-3 monoclonal antibody BMS-986016 IV on days 1 and 15. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive Anti-PD-1 (nivolumab) IV over 60 minutes on days 1 and 15 and urelumab IV on day 1. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.

(2pts enrolled before the Anti-CD137 antibody (BMS-663513 - urelumab) treatment arm closed by BMS on 10/16/18 due to closure of BMS Urelumab development program. Subjects currently on treatment may continue.)

INTRATUMORAL STUDIES: Patients enrolled on the Intratumoral Studies surgical arm pre-operatively receive either anti-LAG-3 monoclonal antibody BMS-986016 as in Part A Arm I, urelumab as in as in Part A Arm II, nivolumab and anti-LAG-3 monoclonal antibody BMS-986016 as in Part B Arm I, or nivolumab and urelumab as in Part B Arm II. Within 45 days of surgical resection, patients post-operatively receive either anti-LAG-3 monoclonal antibody BMS-986016 as in Part A Arm I, urelumab as in as in Part A Arm II, nivolumab and anti-LAG-3 monoclonal antibody BMS-986016 as in Part B Arm I, or nivolumab and urelumab as in Part B Arm II.

(3pts enrolled before the Anti-CD137 antibody (BMS-663513 - urelumab) treatment arm closed by BMS on 10/16/18 due to closure of BMS Urelumab development program. Subjects currently on treatment may continue.)

After completion of study treatment, patients are followed up at 60 days, every 2 months for 2 years, and then every 6 months thereafter. Patients taken off treatment for other reasons than disease progression are followed up every 2 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven glioblastoma or gliosarcoma which is progressive or recurrent following radiation therapy and temozolomide

  * Tumor O-6-methylguanine-deoxyribonucleic acid (DNA) methyltransferase (MGMT) methylation status must be available; results of routinely used methods for MGMT methylation testing (e.g. mutagenically separated polymerase chain reaction [MSPCR] or quantitative polymerase chain reaction [PCR]) are acceptable
  * Patients must have measurable contrast-enhancing disease (defined as at least 1 cm x 1 cm) by magnetic resonance imaging (MRI) imaging within 21 days of starting treatment (patients may have gross total resection, but should have measurable disease post-operatively); patients must be able to undergo MRI of the brain with gadolinium; patients must be maintained on a stable corticosteroid regimen (no increase for 5 days) prior to this baseline MRI
  * Patients must be in first recurrence of glioblastoma following radiation therapy and temozolomide
  * Patients must have recovered from severe toxicity of prior therapy; an interval of at least 12 weeks must have elapsed since the completion of radiation therapy or placement of Gliadel wafers, and at least 6 weeks must have elapsed from the last dose of temozolomide (TMZ); no prior therapies are allowed other than radiation, temozolomide, and Gliadel wafers (placed during the first surgery at diagnosis of GBM)
  * Patients must have a Karnofsky performance status >= 60% (i.e. the patient must be able to care for himself/herself with occasional help from others)
  * Absolute lymphocyte count >= 1000/ul
  * Absolute neutrophil count >= 1,500/ul
  * Platelets >= 100,000/ul
  * Hemoglobin >= 9 g/dl
  * Total bilirubin =< institutional upper limit of normal
  * Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional upper limit of normal
  * Creatinine =< institutional upper limit of normal OR creatinine clearance >= 60 ml/min/1.73m^2 for patients with creatinine levels above institutional normal
  * Activated partial thromboplastin time (APTT) or partial thromboplastin time (PTT) =< 1.5 x institutional upper limit of normal
  * Patients must be able to provide written informed consent
  * Women of childbearing potential must have a negative serum pregnancy test within 24 hours prior to treatment start; women of childbearing potential must agree to use two methods of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study treatment, and through 23 weeks after the last dose of study drug; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and through 31 weeks after the last dose of study drug
  * Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, breast, or bladder; patients with prior malignancies must be disease-free for >= five years

Exclusion Criteria:

* Patients receiving any other investigational agents are ineligible

  * Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to anti-LAG-3, anti-CD137, and anti-PD1 are ineligible; the investigator brochures can be referenced for more information
  * Patients with active or recent history of known or suspected autoimmune disease are ineligible; subjects with type 1 diabetes mellitus, hypothyroidism only requiring hormone replacement, and skin disorders (vitiligo, psoriasis, or alopecia) not requiring systemic treatment, are permitted to enroll
  * Patients with a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days of study entry are ineligible
  * Patients must not be receiving greater than 1 mg dexamethasone/day (or an equivalent amount of an alternative corticosteroid) for at least 1 week prior to treatment start
  * Patients must have no evidence of mass effect and no midline shift
  * Patients must have no evidence of significant hematologic, renal, or hepatic dysfunction; patients with underlying hepatocellular disease should be given careful risk/benefit consideration prior to enrollment; patients with a history of any chronic hepatitis as evidenced by the following are ineligible:

    * Positive test for hepatitis B surface antigen (HBsAg)
    * Positive test for qualitative hepatitis C viral load (by PCR) (Note: subjects with positive hepatitis C antibody and negative quantitative hepatitis C by PCR are eligible; history of resolved hepatitis A virus infection is not an exclusion criterion)
    * History of alcoholic or non-alcoholic steatohepatitis (NASH), auto-immune hepatitis, or previous grade 3-4 drug-related hepatitis, or any form of chronic liver disease
  * Patients must be hepatitis C virus (HCV) negative (by quantitative PCR [qPCR]) and hepatitis B virus core antibody (HBcAb) negative (no prior hepatitis B infection)
  * Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, clinically significant cardiac disease, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, are ineligible
  * Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with these agents
  * Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of anti-LAG-3 monoclonal antibody BMS-986016 as monotherapy as determined by frequency of toxicity | 4 weeks
  The frequency of toxicity will be tabulated by the tested dose or doses using descriptive statistics. The proportion of subjects who experienced grade 3 or above toxicities (as defined by CTCAE v. 5.0 [Common Terminology Criteria for Adverse Events]) will be estimated, along with 95% confidence interval. MTD will be confirmed as the maximum dose level at which ≤ 33% of participants experience a dose-limiting toxicity (DLT).
Maximum tolerated dose (MTD) of anti-CD137 as monotherapy as determined by frequency of toxicity | 4 weeks
  The frequency of toxicity will be tabulated by the tested dose or doses using descriptive statistics. The proportion of subjects who experienced grade 3 or above toxicities (as defined by CTCAE v. 5.0 [Common Terminology Criteria for Adverse Events]) will be estimated, along with 95% confidence interval. MTD will be confirmed as the maximum dose level at which ≤ 33% of participants experience a dose-limiting toxicity (DLT).
MTD of Anti-LAG-3 + Anti-PD-1 as determined by frequency of toxicity | 4 weeks
  The frequency of toxicity will be tabulated by the tested dose or doses using descriptive statistics. The proportion of subjects who experienced grade 3 or above toxicities (as defined by CTCAE v. 5.0 [Common Terminology Criteria for Adverse Events]) will be estimated, along with 95% confidence interval. MTD will be confirmed as the maximum dose level at which ≤ 33% of participants experience a dose-limiting toxicity (DLT).
MTD of Anti-CD137 + Anti-PD-1 as determined by frequency of toxicity | 4 weeks
  The frequency of toxicity will be tabulated by the tested dose or doses using descriptive statistics. The proportion of subjects who experienced grade 3 or above toxicities (as defined by CTCAE v. 5.0 [Common Terminology Criteria for Adverse Events]) will be estimated, along with 95% confidence interval. MTD will be confirmed as the maximum dose level at which ≤ 33% of participants experience a dose-limiting toxicity (DLT).

SECONDARY OUTCOMES:
Overall Survival | 2 years or until time of death, whichever occurs first
  The Kaplan-Meier method will be used to estimate overall survival probability and median time of survival along with a 95% confidence interval.
Progression-free survival rate | 1 year
  To estimate PFS rate at one year, all patients with non-progressive disease and alive at one year will be evaluated by RANO and iRANO at one year to confirm non-progressive status. The proportion of patients who achieve PFS at one year will be estimated along with a 90% confidence interval, assuming underlying binomial distribution.
Overall Response, assessed by RANO and iRANO | up to 2 years
  To estimate an overall tumor response rate: the proportion of patients who have objective partial response or complete response during the course of treatment will be estimated, along with 95% confidence intervals using the exact binomial method regardless of dosage, single or combination treatment.
Overall Response to anti-LAG-3 monoclonal antibody BMS-98601, assessed by RANO and iRANO | up to 2 years
  The proportion of patients who have objective partial response or complete response to anti-LAG-3 monoclonal antibody BMS-98601 during the course of treatment will be estimated per dose level with 95% confidence interval.
Overall Response to anti-CD137 as monotherapy, assessed by RANO and iRANO | up to 2 years
  The proportion of patients who have objective partial response or complete response to anti-CD137 as monotherapy during the course of treatment will be estimated per dose level with 95% confidence interval.
Overall Response to Anti-LAG-3 + Anti-PD-1, assessed by RANO and iRANO | up to 2 years
  The proportion of patients who have objective partial response or complete response to Anti-LAG-3 + Anti-PD-1 combination therapy, during the course of treatment will be estimated per dose level with 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Micheal Lim, MD, Study Chair — Johns Hopkins/ABTC
Locations (11):
- United States (11):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Abrams Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No